CLINICAL TRIAL: NCT03652792
Title: Single-Dose, Randomized, Open-Label, Two-Way Crossover Study to Evaluate the Bioequivalence of Azilsartan Tablets in Chinese Healthy Volunteers
Brief Title: Bioequivalence Study of Azilsartan Tablets in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Collaborators: Zhaoke (Guangzhou) Pharmaceutical Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ZK-HK-AZI-201705
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Bioequivalence of Two Azilsartan Formulations
MeSH Terms: interventions — azilsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Azilsartan (Zhaoke) Under Fasting (Experimental): Subjects will take a single Azilsartan (Zhaoke) 20mg Tablet under fasting condition
  Interventions: Drug: Azilsartan (Zhaoke)
- Azilsartan (Takeda) Under Fasting (Active Comparator): Subjects will take a single Azilva 20mg Tablet under fasting condition
  Interventions: Drug: Azilsartan (Takeda)
- Azilsartan (Zhaoke) Under Fed (Experimental): Subjects will take a single Azilsartan (Zhaoke) 20mg Tablet under fed condition
  Interventions: Drug: Azilsartan (Zhaoke)
- Azilsartan (Takeda) Under Fed (Active Comparator): Subjects will take a single Azilva 20mg Tablet under fed condition
  Interventions: Drug: Azilsartan (Takeda)

INTERVENTIONS:
Drug: Azilsartan (Zhaoke) — Azilsartan 20mg tablets from Zhaoke
  Other Names: Azilsartan
  Arms: Azilsartan (Zhaoke) Under Fasting; Azilsartan (Zhaoke) Under Fed
Drug: Azilsartan (Takeda) — Azilva 20mg tablets from Takeda
  Other Names: Azilva
  Arms: Azilsartan (Takeda) Under Fasting; Azilsartan (Takeda) Under Fed

SUMMARY:
The purpose of this study was to determine the bioequivalence of two azilsartan formulations after administration of single doses to healthy subjects under fasted and fed conditions. These data were to be evaluated statistically to determine if the products meet bioequivalence criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between 18 and 40 (inclusive) years of age.
2. Weight ≥ 50kg and the body mass index (BMI) within the range 19~24kg/m2 (inclusive);
3. Negative urine hCG pregnancy test.
4. Non-lactating women and willing to use appropriate contraceptive methods such as an intrauterine device (IUD), diaphragm with spermicides or abstinence or have a sterile sexual partner (e.g., vasectomy) during the whole study period. Men willing to use an appropriate method of contraception (such as condom with spermicide or use by partner of oral, implantable or injectable contraceptives, IUD, diaphragm, with spermicides) or abstinence or will have a sterile sexual partner during the whole study period;
5. Subjects understand the nature, significance, possible benefits, inconveniences and potential risks before participating in this trial, understood the trial process, and are voluntary to sign the informed consent form and to participate in this trial.

Exclusion Criteria:

1. Subjects who have abnormalities with clinical significance in physical examination, laboratory examinations, 12-lead ECGs, chest X-ray;
2. Subjects with clinically significant history of orthostatic hypotension, chronic gastrointestinal disease (such as gastric ulcer, gastritis, etc.), renal disease (such as nephritis, pyelonephritis, etc.), or cardiovascular, respiratory, neurological, psychotic, haematological, endocrine or other disorders within the past 6 months before randomization or at the discretion of the investigators;
3. Subjects with allergic history to Angiotensin Receptor Blockers or other anti-hypertensive drugs or anti-hypertensive biological agents;
4. Sitting systolic blood pressure (SBP) <80mmHg or >140mmHg, and/or sitting diastolic blood pressure (DBP) <50mmHg or >90mmHg at screening;
5. With the history of using any drug which will inhibit (chlorpromazine, cimetidine, ciprofloxacin, metronidazole, chloramphenicol, isoniazid and sulphonamide) or induce liver metabolize drug (barbiturate, carbamazepine, aminoglutethimide, grifulvin, ethanol, ammonia methyl propyl, phenytoin, rifampin, glutethimide, dexamethasone, sulfinpyrazone) within 1 month before randomization;
6. Vegetarian or abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits within the past 4 weeks prior to screening;
7. History of alcohol abuse in the last 6 months prior to screening defined as an average weekly intake of greater than 14 unit (one unit is equivalent to 360ml of beer or 45ml of spirits with 40% alcohol content or 150 ml of wine); or subjects with positive alcohol breath test;
8. History of smoking >5 cigarettes a day in the last 6 months prior to screening;
9. History of drug abuse and taking drugs (such as marijuana, cocaine, opiates, benzodiazepines, amphetamines, barbiturates, tricyclic antidepressant) or subjects with positive urine drug abuse test results;
10. Consumption of excessive amount of tea, coffee and/or caffeinated beverage (more than 8 cups/day, 200mL/cup) in the last 1 month prior to screening;
11. Subjects who have participated in clinical trial (as subjects) in the last 3 months prior to screening;
12. Blood donation of 250 ml or more in the 3 months prior to screening;
13. Positive result of hepatitis B antigen, hepatitis C antibody, HIV antibody or syphilis antibody;
14. Consumption of grapefruit juice, xanthine diet, chocolate, coffee or tea, carbonated beverages, or any other caffeinated beverages within 48 hours before randomization;
15. Strenuous exercise within 48 hours before randomization;
16. Administered any drugs (prescription medicine, over-the-counter drug, vitamins, supplements and Chinese herbal medicine) within 2 week before randomization; topical treatment is generally allowed or based on investigators' judgement.
17. Subjects who, in the opinion of the investigators, should not participate in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
Bioequivalence under Fasting Condition | 48 hours
Bioequivalence under Fed Condition | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Phase I Clinical Trial Centre, Chinese University of Hong Kong, Hong Kong, Sha Tin New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No